CLINICAL TRIAL: NCT00115622
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Study to Evaluate the Efficacy and Safety of Once-Daily, Intranasal Administration of GW685698X Aqueous Nasal Spray 100mcg for 14 Days in Adult and Adolescent Subjects With Seasonal Allergic Rhinitis
Brief Title: Study In Adults And Adolescents With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR30003
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Hayfever; Rhinitis, Allergic, Seasonal; Seasonal Allergic Rhinitis
Keywords: GW685698X; once daily; mountain cedar; allergic rhinitis; fluticasone furoate
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — fluticasone furoate

INTERVENTIONS:
Drug: fluticasone furoate

SUMMARY:
The purpose of the study is to compare the efficacy and safety of an investigational nasal spray compared with placebo nasal spray in the treatment of seasonal allergic rhinitis. Allergic rhinitis is an inflammatory disorder of the upper airway that occurs following allergen exposure. The focus of this study, seasonal allergic rhinitis (SAR), is one type of allergic rhinitis that is triggered by the pollen from trees, grasses, and weeds. Commonly referred to as "hay fever", it is characterized by sneezing, nasal congestion and pruritus, rhinorrhea, and pruritic, watery, red eyes.

ELIGIBILITY:
Inclusion criteria:

* Informed consent.
* Outpatient.
* Females must use appropriate contraception.
* Diagnosis of seasonal allergic rhinitis.
* Adequate exposure to allergen.
* Able to comply with study procedures.
* Literate.

Exclusion criteria:

* Significant concomitant medical condition.
* Use of corticosteroids, allergy medications, or tobacco.
* Clinically significant abnormal ECG.
* Laboratory abnormality.
* Positive pregnancy test.
* Allergy to any component of the investigational product.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2004-12; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline over the entire treatment period in daily, reflective, total nasal symptom scores.
Mean change from baseline over the entire treatment period in the daily, reflective, total ocular symptom score.

SECONDARY OUTCOMES:
Mean change from baseline over the entire treatment period in AM, pre-dose, instantaneous, total nasal symptom score.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, New Braunfels, Texas
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Hampel FC Jr, Jacobs R, Martin B. Toler T, Ellsworth A, Philpot E. Once-daily fluticasone furoate* nasal spray (FF) provides 24-hour symptom relief in subjects with seasonal allergic rhinitis (SAR) caused by mountain cedar pollen. *USAN approved name. J
- [Background] Jacobs R, Martin B, Hampel F, Toler W, Ellsworth A, Philpot E. Effectiveness of fluticasone furoate 110 microg once daily in the treatment of nasal and ocular symptoms of seasonal allergic rhinitis in adults and adolescents sensitized to mountain cedar pollen. Curr Med Res Opin. 2009 Jun;25(6):1393-401. doi: 10.1185/03007990902890512. PMID 19419338
- [Background] Ratner P, Andrews C, van Bavel J, Toler T, Ellsworth A, Philpot E. Once-daily fluticasone furoate* nasal spray (FF) effectively treats ocular symptoms of seasonal allergic rhinitis (SAR) caused by mountain cedar pollen. *USAN approved name. J Allergy Cli
- [Background] van Bavel J, Toler T, Ellsworth A, Stanford R, Philpot E. Once-daily fluticasone furoate* nasal spray (FFNS) improves quality of life (QoL) in subjects with seasonal allergic rhinitis (SAR) during the mountain cedar pollen season. *USAN approved name. J
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: FFR30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR30003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register